CLINICAL TRIAL: NCT05520476
Title: Neuroliten MVP System Clinical Observation Study
Status: Active, not recruiting | Type: Observational
Sponsor: Enliten AI (Industry)
Collaborators: CSSi Life Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: EL-001
Record Dates: First submitted 2022-08-23; First posted 2022-08-30 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy
Keywords: Seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 20 patients with at least two seizures per week.: The device collects vital signs and EEG data as well as caregiver information associated with seizure episodes.
  Interventions: Device: Neuroliten MVP system

INTERVENTIONS:
Device: Neuroliten MVP system — The Neuroliten MVP system will be an App that gets uploaded to the patients iPhone from the App Store.

SUMMARY:
This is an observational study for data collection from subjects diagnosed with Epilepsy/intractable seizures. The Neuroliten MVP System will not be used for patient management or treatment decisions.

DETAILED DESCRIPTION:
Neuroliten MVP system stores the data obtained from wearables, caregivers, and all audio/video recording of seizure activity that the caregiver captures associated with a seizure episode.

The primary objective of this study is to obtain vital signs and neurological indicators via the Neuroliten MVP System to correlate to the onset of seizures that are detected by the observations of family/caregivers.

The secondary objective is to identify the vital signs and/or neurological indicators that are associated with seizure onset.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) approved informed consent is signed and dated before any study-related activities.
2. Male and female subjects ages 18 to 75, inclusive.
3. Documented history of at least two (2) seizures per week. Seizures can be generalized and/or focal.
4. Diagnosed with intractable or refractory epilepsy.
5. Have a caregiver/family member who stays with the subject, has the ability to detect seizures, and is willing to provide the information needed for the study.
6. Have implanted vagus nerve stimulation (VNS).
7. Have the ability to understand the requirements of the study and are willing to comply with all study requirements.
8. Must have a working Apple iPhone.

Exclusion Criteria:

1. Women who are either pregnant or breastfeeding.
2. Subjects unable/unwilling to wear the Apple Watch and EEG Wearable for extended periods.
3. Requires the use of a ventilator.
4. Requires the use of supplemental oxygen.
5. Uses a pacemaker or other electronic neurostimulator, except the VNS.
6. Any medical or surgical condition that in the opinion of the investigator may interfere with participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a documented history of at least 2 seizures per week.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | 90 days
  Heart Rate (beats per minute)
Oxygen Saturation | 90 days
  Oxygen Saturation (SpO2 %)
Respiratory Rate | 90 days
  Respiratory Rate (breaths per minute)
Blood Pressure | 90 days
  Blood Pressure (mmHg)
Temperature | 90 days
  Temperature (Fahrenheit)
Brain Signals | 90 Days
  Brain signals obtained using a 14-channel EEG Wearable

SECONDARY OUTCOMES:
Clinical Observations from Caregiver | 90 days
  Caregiver will log details of specific seizure episodes with the following measures:
  * Date, Time and Duration of Seizure
  * Type of seizure (if known)
  * Caregiver's assessment of severity (1-10, 10 being very severe)
  * Cluster of seizures (How many were observed and interval)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hager, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Loveland, Colorado, United States

IPD SHARING:
Plan to Share IPD: No